CLINICAL TRIAL: NCT03959280
Title: Tailored Intervention on Nutrition and Exercise for Obstructive Sleep Apnea Patients Treated With CPAP
Brief Title: CPAP, Nutrition & Exercise Against Sleep Apnea
Acronym: TINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Raphael Heinzer (Other)
Collaborators: Swiss Lung Association (Unknown); Ligue Pulmonaire Vaudoise (Unknown)
Responsible Party: Sponsor-Investigator, Raphael Heinzer, Prof., Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00586
Record Dates: First submitted 2019-05-14; First posted 2019-05-22 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Sleep Apnea; Overweight and Obesity
Keywords: obstructive sleep apnea; CPAP therapy; exercise; diet; quality of life
MeSH Terms: conditions — Sleep Apnea Syndromes; Overweight; Obesity; Sleep Apnea, Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored intervention (Experimental): In this group, participants will receive a comprehensive lifestyle program in addition to CPAP therapy which will include a supervised exercise program, diet interventions and behavioural counselling during 12 weeks.
  Then, participants will follow a real-world maintenance program from weeks 12 to 24. It will include one telephone-based contact per month with the study coordinator. Participants will be encouraged to maintain their lifestyle modification during this phase.
  Interventions: Other: Tailored intervention
- Control (Active Comparator): Participant in this group will benefit from routine CPAP therapy management from week 0 to 24.
  Interventions: Other: Control

INTERVENTIONS:
Other: Tailored intervention — * The exercise program consists of 2 x 1.5-hour supervised nordic walking sessions weekly during 12 weeks and 1-hour unsupervised moderate physical activity per week from week 4.
  * The diet intervention includes one face-to-face consultation with a dietician and one telephone-based contact monthly, i.e. 6 diet interventions for 12 weeks.
  * Behavioural changes techniques will be included in diet and exercise interventions.
  Other Names: TINE
  Arms: Tailored intervention
Other: Control — This intervention will include tailored instruction on CPAP use and standard advices on physical activity and nutrition at CPAP initiation.
  Other Names: CPAP
  Arms: Control

SUMMARY:
This study evaluates the addition of a comprehensive lifestyle program including dietary management and exercise to continuous positive airway pressure (CPAP) therapy in overweighted adults with obstructive sleep apnea. Half of the participants will receive CPAP therapy while the other half will have diet consultations, nordic walking sessions and CPAP.

DETAILED DESCRIPTION:
While the specific impact of obstructive sleep apnea (OSA) on quality of life is well established, the impact of CPAP therapy on quality of life remains unclear. Yet, improving the quality of life of OSA patient is one of the main targets of treatment.

Both exercise and healthy diet are recommended in the management of overweight and obesity. This should improve quality of life as well as comorbidities associated with sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed for obstructive sleep apnea and requiring CPAP therapy
* BMI>25and≤40kg/m2
* Low physical activity (< 150 min of MVPA per week)
* IAH≥15
* Able to give informed consent as documented by signature

Exclusion Criteria:

* Patients already treated for OSA or another sleep disorder
* Required use of supplemental oxygen
* Active infection, malignancy or chronic inflammatory disorders
* More than moderate alcohol use of > 14 drinks per week
* Severe depression defined by a BDI > 30
* Surgery within the previous 3 months
* Known cardiac or pulmonary disease contraindicating exercise training
* Patient with a bariatric surgery project or already operated
* Pregnant or lactating women
* Onset of a severe cardiac disease contraindicating exercise training
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, peripheral functional limitation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life: SF-36 | 12 weeks
  Mean difference in the general health perception (GH) domain on the Medical Outcome Study Short Form (SF-36) between groups

SECONDARY OUTCOMES:
General quality of life: SF-36 | 12 and 24 weeks
  Mean difference in the seven other following SF-36 subscales between groups:
  * Vitality (VT)
  * physical functioning (PF)
  * bodily pain (BP)
  * Role-physical (RP)
  * Role-emotionale (RE)
  * Social functioning (SF)
  * Mental health (MH)
  Each subscale ranges from 0 to 100. The higher the score, the better quality of life.
Specific quality of life: Calgary Sleep Apnea Quality of Life Index (SAQLI) | 12 and 24 weeks
  Mean difference in the SAQLI global score and score in the domain A, B, C and D between groups.
  The SAQLI is a 35-items instrument that captures the adverse impact of sleep apnea on 4 domains:
  * Daily functioning (A)
  * Social interactions (B)
  * Emotional functioning (C)
  * Symptoms (D)
  When the SAQLI is administered after a therapeutic intervention, a fifth domain (E) is completed (Treatment-related symptoms).
  Items are scored on a 7-point scale with "all of the time" and "not at all" being the most extreme responses. Item and domain scores are averaged to yield a composite total score between 1 and 7. Higher scores represent better quality of life.
  To obtain the global SAQLI score the sum of the mean domain scores A, B, C, and D is divided by 4. If Domain E has been used after a therapeutic intervention, the SAQLI score is obtained by summing the mean domain scores A, B, C, and D, subtracting the mean Domain E score and dividing by 4.
Daytime excessive sleepiness | 12 and 24 weeks
  Mean difference in the Epworth Sleepiness Scale (ESS) score between groups. The ESS is a 8-item questionnaire. ESS score can range from 0 to 24. The higher the ESS score, the higher daytime sleepiness.
Subjective sleep quality | 12 and 24 weeks
  Mean difference in the Pittsburgh Sleep Quality Index (PSQI) score between groups.
  The PSQI is a 19-item questionnaire which measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by summing the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Mood | 12 and 24 weeks
  Mean difference in the Hospital Anxiety Depression Scale (HADS) score between groups.
  The HADS is a 14-item questionnaire. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3. Scores range from 0 to 21 for either anxiety or depression. The higher the scores, the more anxiety and depression symptoms are important.
Depression | 12 and 24 weeks
  Mean difference in the Beck depression inventory (BDI) score between groups. The BDI is a 21-item questionnaire which assess the severity of depression. Score range from 0 to 63. Higher values represent a worse outcome.
Fatigue | 12 and 24 weeks
  Mean difference in the Pichot scale score between groups. The Pichot Scale is a 8-item questionnaire to assess fatigue. The score ranges from 0 to 32. Higher score indicates greater fatigue.
Blood pressure | 12 and 24 weeks
  Mean difference in systolic and diastolic blood pressure measured at office as well as via a 24-h ambulatory blood pressure monitoring
Weight | 12 and 24 weeks
  Mean difference in weight (kg) between groups
Height | 12 and 24 weeks
  Mean difference in height (m) between groups
Body-mass index (BMI) | 12 and 24 weeks
  Mean difference in BMI (kg.m^2) between groups. Weight will be divided by the square of the height to report BMI in kg/m^2.
Waist circumference | 12 and 24 weeks
  Mean difference in waist size (cm) between groups
Hip circumference | 12 and 24 weeks
  Mean difference in hip size (cm) between groups
Waist-hip ratio | 12 and 24 weeks
  Mean difference in waist/hip ratio between groups
Neck size | 12 and 24 weeks
  Mean difference in neck circumference (cm) between groups
Fat distribution | 12 and 24 weeks
  Mean difference in fat-free mass and fat mass measured via bioimpedance analysis between groups
Resting metabolism | 12 and 24 weeks
  Mean difference in basal metabolic rate (BMR) between groups using indirect calorimetry
Concentration of fasting glucose | 12 and 24 weeks
  Mean difference in fasting glucose (mg/dL) between groups
Rate of glycosylated haemoglobin | 12 and 24 weeks
  Mean difference in glycosylated haemoglobin [HbA1c] (%) between groups
Concentration of insulin | 12 and 24 weeks
  Mean difference in insulin (mlU/L) between groups
Concentration of total cholesterol | 12 and 24 weeks
  Mean difference in total cholesterol (g/L) between groups
Concentration of HDL cholesterol | 12 and 24 weeks
  Mean difference in HDL cholesterol (g/L) between groups
Concentration of LDL cholesterol | 12 and 24 weeks
  Mean difference in LDL cholesterol (g/L) between groups
Concentration of triglycerides | 12 and 24 weeks
  Mean difference in triglycerides (g/L) between groups
Concentration of ultrasensible CRP | 12 and 24 weeks
  Mean difference in CRP-US (mg/L) between groups
Respiratory events | 12 and 24 weeks
  Mean difference in apnea-hypopnea index (AHI) during sleep between groups measured via ambulatory polygraphy
Desaturation events | 12 and 24 weeks
  Mean difference in oxygen desaturation index (ODI) during sleep between groups measured via ambulatory polygraphy
T90% | 12 and 24 weeks
  Mean difference in percentage time spent with an oxygen saturation (SpO2) < 90% (T90%) during sleep between groups using an oximeter.
Nocturnal hypoxic load | 12 and 24 weeks
  Mean difference in hypoxic load related to apnea-hypopnea events and to sleep stages between groups using an ambulatory polygraphy. The area under the desaturation curve (SpO2) associated with respiratory-events will be used to quantify the 'hypoxic load'.
Autonomic Arousal Index (Aai) | 12 and 24 weeks
  Mean difference in pulse wave amplitude (PWA) drop during sleep between groups using an ambulatory polygraphy
Autonomic Arousal Area under the curve | 12 and 24 weeks
  Mean difference in the sum of the autonomic arousal area under the curve (AUC) between groups using an ambulatory polygraphy
Autonomic Arousal duration | 12 and 24 weeks
  Mean difference in the sum of the duration of the PWA drops between groups using an ambulatory polygraphy
CPAP withdrawal | 12 and 24 weeks
  Proportion of CPAP withdrawal in each arms
CPAP adherence | 12 and 24 weeks
  Mean duration of CPAP use per night in each arms
CPAP compliance | 12 and 24 weeks
  Proportion of compliant patients (mean CPAP use > 4h per night) in each arm
Medical visit | 12 and 24 weeks
  Mean number of medical visits between groups
Sedentary behaviour | 12 and 24 weeks
  Mean difference in sedentary time (min per day) between groups using accelerometer
Light physical activity (LPA) behaviour | 12 and 24 weeks
  Mean difference in LPA time (min per day) between groups using accelerometer
Moderate to vigorous physical activity | 12 and 24 weeks
  Mean difference in MVPA (METs-min per week) between groups using accelerometer
Exercise capacity | 12 and 24 weeks
  Mean difference in the distance (m) on the incremental shuttle walking test (ISWT) between groups
Postural stability | 12 and 24 weeks
  Mean difference in balance stability (total displacement of the centre of pressure) between groups using a posturographic platform

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Heinzer, MD, PhD, Principal Investigator — University Hospital of Lausanne, Switzerland
Locations (2):
- Centre Hospitalier Universitaire Saint-Etienne, Saint-Etienne, France
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the Ligue Pulmonaire Vaudoise — https://www.liguepulmonaire.ch/fr/ligue-pulmonaire-vaudoise/page-daccueil.html